CLINICAL TRIAL: NCT03965897
Title: Preventing Persistent Post-Surgical Pain and Dysfunction in At-Risk Veterans: Effect of a Brief Behavioral Intervention
Brief Title: Preventing Persistent Post-Surgical Pain and Dysfunction
Acronym: PrePARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara A Rakel (Other)
Collaborators: Baylor College of Medicine (Other); National Institute of Nursing Research (NINR) (NIH); Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Barbara A Rakel, Professor and Associate Dean of Research, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201812794; 1R01NR017610-01A1 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pain; Function; Anxiety; Depression; Arthroplasty, Replacement, Knee; Veterans
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study uses a cluster randomization approach where the unit of randomization is the workshops. Randomization occurs at the start of each workshop so that all participants attending that workshop are randomized to that intervention (i.e. ACT vs. AC). Statistician Dr. Zimmerman generates the randomization sequence using PLAN procedure (SAS v9.2). Randomization of workshops occurs in permuted blocks of 2 and 4 and are stratified by site (i.e. Iowa City versus Houston).
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study. Participants and outcome assessors are blinded to treatment. Allocation to intervention group remains concealed until the beginning of the workshop when all invited participants have arrived. Those in attendance will receive the assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention Control (AC) (Active Comparator): The primary purpose of this workshop is to provide attention and education to participants. Topics of discussion will include: a) the pathophysiology of postoperative pain and how it differs from preoperative pain, b) the role of contextual factors (e.g., depressive or anxiety symptoms, expectation) on the experience of pain, d) the role of inflammation in pain and healing, e) types of pain medications and other pain relief strategies provided following surgery, and f) goals of pain medications. Additionally, deep (diaphragmatic) breathing strategies will be taught and a progressive muscle relaxation exercise will be performed in the workshop at strategic times to maintain Veteran engagement.
  Interventions: Other: Attention Control (AC)
- Acceptance and Commitment Therapy (ACT) (Experimental): The ACT intervention will include: 1) Acceptance and Mindfulness Training emphasizing new ways of managing troubling thoughts, feelings, and physical sensations (e.g., learning how to recognize, and develop cognitive distance from, unhelpful thoughts such as "I can't take this pain anymore" or "This is unfair") and learning how to willingly face experiences that cannot be changed; and 2) Behavioral Change Training involving a) teaching patients how to recognize ineffective patterns of behavior and habits, b) exploring and setting life goals and goals related to mental and physical health, and c) promoting effective and committed actions to achieve these goals despite the urge to do otherwise. The workshop will also include information on pain and pain control post-TKA.
  Interventions: Behavioral: Acceptance and Committment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Committment Therapy (ACT) — Overall, the goal of the ACT intervention is to cultivate psychological flexibility: to help Veterans respond to life events in ways which do not exacerbate difficulties or restrict engagement in meaningful activities. It increases patients' awareness of behaviors that exacerbate the pain (such as struggling with it) and recognition of avoidance strategies that interfere with life engagement.
  Arms: Acceptance and Commitment Therapy (ACT)
Other: Attention Control (AC) — Information on any other coping practices will be omitted. The group facilitators will present one topic at a time, using the Pain Manual, and the participants will discuss and reflect about issues and experiences related to each topic. If necessary, the group facilitators will raise specific discussion questions to facilitate group dialogue and participant involvement.
  Arms: Attention Control (AC)

SUMMARY:
Primary Aim: To examine the superior efficacy of ACT versus Attention Control (AC) on postoperative pain intensity and functioning in at-risk Veterans undergoing TKA. Changes in pain intensity and functioning from baseline to 6 weeks, 3 months and 6 months post-TKA will be compared. Level of pain intensity will be measured using the BPI Pain Severity Subscale and level of functioning will be measured using the KOOS Activities of Daily Living and Quality Of Life Subscales.

Secondary Aims: A) To examine the superior efficacy of ACT versus AC on the severity of anxiety and depressive symptoms and improvements in coping skills. Changes from baseline to 6 weeks, 3 months and 6 months post-TKA will be compared. Anxiety and depressive symptoms will be measured with the Hamilton Rating Scales (Ham-A and Ham-D, respectively). Coping skills (i.e. Pain Acceptance and Engagement in Values-Based Behavior) will be measured with the Chronic Pain Acceptance Questionnaire and the Chronic Pain Values Inventory. B) To evaluate whether decreases in distress-based symptoms and increases in coping skills mediate changes in pain and functioning at 6 months in Veterans receiving ACT. Changes in anxiety symptoms, depressive symptoms, pain acceptance and engagement in values-based behavior from baseline to 6 weeks and 3 months will be used as potential mediators for changes in pain and functioning at 6 months.

Exploratory Aim: Describe the pharmacological and non-pharmacological strategies Veterans are using to manage pain and their perceived helpfulness. This will provide insights into the effects of the current opioid restrictions on pain management strategies. These strategies & their perceived helpfulness will be assessed using the Pain Management Strategies Survey at baseline, 6 weeks, 3, and 6 months.

DETAILED DESCRIPTION:
Persistent post-surgical pain (PPSP) is a common and debilitating problem following surgery.1 Orthopedic surgeries, such as Total Knee Arthoplasty (TKA), are consistently associated with high postoperative pain, putting patients at risk for PPSP.2, 3 In fact, TKA has the highest rate of PPSP at 6 months (49%) when compared to a variety of surgeries.4 Pain that persists beyond the expected period of healing serves little or no useful purpose and can be devastating to one's sense of well-being. Notably, pain severity is highly correlated with adverse effects on physical functioning, recovery and quality of life, including negative impacts on sleep, mood, daily activities, cognitive functions and social life.2, 5-13 PPSP is also highly correlated with prolonged opioid use following surgery. When pain and addiction are present, the patient's level of desperation rises, medical and psychiatric illness severity increases, and there is greater utilization of health care services.

Strong and consistent evidence indicates that patients with high levels of pain, anxiety and/or depressive symptoms (distress) prior to surgery are at risk for PPSP.5, 14-23 Notably, Veterans are at a particularly high risk for post-surgical problems because 80% experience some level of psychological distress prior to surgery and 50% report experiencing pain on a regular basis.9, 24 Furthermore, surgery presents a unique set of circumstances in which the precise timing of the physical insult and ensuing pain are known in advance. 25 It is, therefore, possible and critical that these risk factors be attended to in order to improve postoperative pain management and disrupt processes responsible for the transition from acute to chronic pain.

As proof of concept, co-PIs Rakel and Dindo completed an R34-funded study evaluating the feasibility and potential efficacy of an intensive 1-day Acceptance and Commitment Therapy (ACT) workshop for preventing PPSP and prolonged opioid use following orthopedic surgery in at-risk Veterans. ACT is trans-diagnostic, with effectiveness across a range of conditions, including chronic pain, depression, and anxiety.16-18 The brief, 1-day format was used to optimize treatment adherence and chances for dissemination into clinical settings. Results were promising. 100% of the Veterans attending, completed the 1-day intervention. Compared to controls, Veterans randomly assigned to ACT reported a larger decrease in pain intensity 3 months post-TKA and reached pain and opioid cessation criteria sooner. Importantly, Veterans reporting larger changes in behavioral engagement (targeted mediator of ACT) exhibited significantly larger decreases in pain and opioid use. This application builds on these promising preliminary findings using a rigorous design to establish the unique effects of ACT beyond attention and explore mediators of treatment response.

In the context of the current opioid epidemic, it is also important for us to better understand how changes in opioid prescribing patterns are influencing postoperative pain management strategies. It is likely that complaints of pain will increase, putting patients at higher risk for PPSP and impaired functioning. Early reports suggests that patients are looking for substitute sources of pain relief, such as rogue Fentanyl powder and Gabapentin.26, 27 Using a multi-site, double-blind, two-arm, parallel, randomized controlled trial with Veterans at-risk for PPSP post-TKA, the following aims will be addressed:

Primary Aim: To examine the superior efficacy of ACT versus Attention Control (AC) on postoperative pain intensity and functioning in at-risk Veterans undergoing TKA. Changes in pain intensity and functioning from baseline to 6 weeks, 3 months and 6 months post-TKA will be compared. Level of pain intensity will be measured using the BPI Pain Severity Subscale and level of functioning will be measured using the KOOS Activities of Daily Living and Quality Of Life Subscales.

Secondary Aims: A) To examine the superior efficacy of ACT versus AC on the severity of anxiety and depressive symptoms and improvements in coping skills. Changes from baseline to 6 weeks, 3 months and 6 months post-TKA will be compared. Anxiety and depressive symptoms will be measured with the Hamilton Rating Scales (Ham-A and Ham-D, respectively). Coping skills (i.e. Pain Acceptance and Engagement in Values-Based Behavior) will be measured with the Chronic Pain Acceptance Questionnaire and the Chronic Pain Values Inventory. B) To evaluate whether decreases in distress-based symptoms and increases in coping skills mediate changes in pain and functioning at 6 months in Veterans receiving ACT. Changes in anxiety symptoms, depressive symptoms, pain acceptance and engagement in values-based behavior from baseline to 6 weeks and 3 months will be used as potential mediators for changes in pain and functioning at 6 months.

Exploratory Aim: Describe the pharmacological and non-pharmacological strategies Veterans are using to manage pain and their perceived helpfulness. This will provide insights into the effects of the current opioid restrictions on pain management strategies. These strategies & their perceived helpfulness will be assessed using the Pain Management Strategies Survey at baseline, 6 weeks, 3, and 6 months.

This project builds on promising preliminary data and has the potential to translate what is known about effective treatments of chronic pain to prevent poor surgical outcomes. It incorporates an interdisciplinary approach to the care of Veterans that attends to major risk factors of postoperative sequelae that significantly impact Veterans' quality of life and healthcare utilization. Using an effective, highly accepted and deployable intervention increases the clinical usefulness of these results which may be extended in the future to the many other conditions leading to chronic pain in both Veterans and Civilians.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for unilateral total knee arthroplasty (TKA)
* identified to be "at-risk" at the enrollment visit (i.e. worst pain ≥7 on BPI (severe pain) OR worst pain ≥3 (moderate pain) on BPI PLUS anxiety symptoms ≥6 on the Anxiety Subscale of the Depression, Anxiety and Stress Scale [DASS-21] or ≥10 on the Stress Subscale of the Depression, Anxiety and Stress Scale [DASS-21] OR depressive symptoms ≥7 on Depression Subscale of the Depression, Anxiety and Stress Scale [DASS-21] OR >20 on the Pain Catastrophizing Scale [PCS].

Exclusion Criteria:

* inability to complete study forms/procedures because of a language/literacy barrier;
* bipolar or psychotic disorder
* history of brain injury
* cognitive impairment (determined by score of <21 [high school or above] or <20 [< high school] on the Veterans Affairs Saint Louis University Mental Status [SLUMS] exam)
* ACT therapy within the past year
* inability to attend workshop prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (preop) to 6 months post-surgery.
  Pain will be measured using the Brief Pain Inventory (BPI) Short Form.
Function | Baseline (preop) to 6 months post-surgery
  Functioning will be measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS).

SECONDARY OUTCOMES:
Anxiety | Baseline (preop) to 6 months post-surgery
  Anxiety will be measured using the Anxiety Subscale of the Depression, Anxiety and Stress Scale (DASS-21).
Depressive Symptoms | Baseline (preop) to 6 months post-surgery
  Depressive Symptoms will be measured using the Depression Subscale of the Depression, Anxiety and Stress Scale (DASS-21).
Level of Pain Acceptance | Baseline (preop) to 6 months post-surgery
  Pain Acceptance will be measured using the Chronic Pain Acceptance Questionnaire (CPAQ).
Level of Success in Engagement in Values-Based Behavior | Baseline (preop) to 6 months post-surgery
  Engagement in Values-Based Behavior will be measured using the Chronic Pain Values Inventory (CPVI).
Pain Management Strategies used | Baseline (preop) to 6 months post-surgery
  Pain Management Strategies will be measured using a Pain Management Strategies Survey (PMSS).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rakel, PhD, Principal Investigator — University of Iowa
Locations (1):
- Iowa City VAMC, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Shanahan ML, Zimmerman B, Rodrigues M, Green D, Embree J, Buckwalter J, Garvin L, Hadlandsmyth K, Smith T, Rakel B, Dindo L. Intersectional pain disparities and resilience in veterans with chronic pain. Health Psychol. 2026 Jan;45(1):123-135. doi: 10.1037/hea0001555. PMID 41396638
- [Derived] Dindo L, Hadlandsmyth K, Garvin L, Marchman J, Zimmerman MB, Buckwalter JA 4th, Green DM, Wollaeger JK, Strayer A, Kim KS, Liu W, Embree J, Rodrigues M, Rakel BA. ACT for postsurgical pain and dysfunction in at-risk veterans: Multisite, double-blind, cluster RCT. J Psychosom Res. 2025 Nov;198:112393. doi: 10.1016/j.jpsychores.2025.112393. Epub 2025 Sep 24. PMID 41032959